CLINICAL TRIAL: NCT00350675
Title: Medical Utilization, Psychotropic Prescriptions, and Somatic Complaints in Israel During the Second Intifada: An Ecological Study of the Impact of Stress.
Brief Title: Medical Utilization in Israel During Second Intifada
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-06-4194-RG-CTIL
Record Dates: First submitted 2006-07-09; First posted 2006-07-11 (Estimated); Last update posted 2006-07-11 (Estimated); Status verified 2006-07

CONDITIONS: Anxiety; Depression; Stress
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
In this ecological study we examine the impact of stress from repeated terrorist attacks during the second initifada on medical utilization by the Israeli population. We hypothesize that in weeks following serious terror attacks there will be an increase in prescriptions for psychiatric medications and an increased number of unexplained somatic complaints. We will also examine associations with overall medical utlization. We will consider age, gender and effects of geographic poximity to location of attacks.

ELIGIBILITY:
Inclusion Criteria:

Ecological study We will examine patterns of visits and prescirptions for all participants in two large health provider institutions in Israel.

Exclusion Criteria:

None - ecological study

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Lipsitz, PhD, Principal Investigator — Gertner Institute, Sheba Medical Center; Raz Gross, MD, Study Chair — Gertner Institute, Sheba Medical Center